CLINICAL TRIAL: NCT05320588
Title: A Phase 1/2 Study of BIO-106 As Monotherapy or In Combination With Pembrolizumab in Patients With Advanced Cancers (StarBridge-1)
Brief Title: A Study in Patients With Advanced Cancers
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BiOneCure Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: StarBridge-1
Record Dates: First submitted 2022-04-02; First posted 2022-04-11 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Advanced Cancer; Advanced Solid Tumor; Cancer; Oncology
MeSH Terms: conditions — Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Multiple ascending dose and dose-expansion of BIO-106 administered as a single agent or in combination with pembrolizumab.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single agent BIO-106 (Experimental): Escalating doses followed by expansion targeting advanced cancers
  Interventions: Drug: BIO-106
- Combination BIO-106 plus pembrolizumab (Experimental): Escalating doses followed by expansion targeting advanced cancers
  Interventions: Drug: BIO-106; Drug: Pembrolizumab

INTERVENTIONS:
Drug: BIO-106 — BIO-106 is a novel antibody-drug conjugate (ADC) that targets the human trophoblast cell surface antigen 2 (Trop-2)
Drug: Pembrolizumab — Programmed death receptor-1 (PD 1)-blocking antibody
  Other Names: Keytruda
  Arms: Combination BIO-106 plus pembrolizumab

SUMMARY:
A first-in-human study using BIO-106 as a single agent and in combination with pembrolizumab in advanced cancers.

DETAILED DESCRIPTION:
This is an open-label, Phase 1/2, first-in-human (FIH), multiple ascending dose and dose-expansion study of BIO-106 administered as monotherapy and in combination with pembrolizumab. Phase 1 will define the maximum tolerated dose (MTD) or recommended Phase 2 dose (RP2D) of BIO-106 that can be advanced to Phase 2. Phase 2 will define the preliminary efficacy of these regimens in the setting of advanced solid tumors with high unmet medical needs.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients histologically or cytologically documented, locally advanced or metastatic solid tumor.
* Disease progression confirmed by imaging or other objective evidence after having received standard treatment; or patients with refractory solid tumors who cannot tolerate standard treatment or have contraindications to standard treatment.
* Measurable disease as determined by RECIST v.1.1 or bone only disease.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Key Exclusion Criteria:

* History of severe hypersensitivity to any ingredient of the study drug(s), including pembrolizumab or other monoclonal antibody.

Impaired cardiac function or history of clinically significant cardiac disease

* Human Immunodeficiency virus (HIV) infection, active hepatitis B infection, or hepatitis C infection.
* Active SARS-CoV-2 infection.
* Untreated central nervous system (CNS), epidural tumor or metastasis, or brain metastasis.

Other protocol defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Estimated)
Dates: Start 2022-03-25 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) and serious adverse events (SAEs) - (Phase 1) | 1 year
  Escalation period
Incidence and nature of dose-limiting toxicities (DLTs) - (Phase 1) | up to 21 days
  Escalation period
Maximum tolerable dose (MTD) or a tolerated dose below MTD - (Phase 1) | 1 year
  Escalation period
Anti-tumor activity by objective response rate (ORR), disease control rate (DCR), duration of response (DOR), progression-free survival (PFS), and overall survival (OS) - (Phase 2) | 2 years
  Expansion period

SECONDARY OUTCOMES:
Anti-tumor activity by objective response rate (ORR), disease control rate (DCR), duration of response (DOR), progression-free survival (PFS), and overall survival (OS) - (Phase 1) | 1 year
  Escalation Period
Incidence of adverse event of special interest (AESI) - (Phase 2) | 2 years
  Expansion period
Incidence of adverse events (AEs) and serious adverse events (SAEs) - (Phase 2) | 2 years
  Expansion period
PK (Cmax) of BIO-106 - (Phase 1/2) | 2 years
  Escalation and expansion periods
PK (AUC) of BIO-106 - (Phase 1/2) | 2 years
  Escalation and expansion periods
Incidence of anti-BIO-106 antibodies - (Phase 1/2) | 2 years
  Escalation and expansion periods

CONTACTS AND LOCATIONS:
Overall Officials: BiOneCure Clinical Development, Study Director — BiOneCure Therapeutics Inc.
Locations (3):
- United States (3):
  - NEXT Oncology Austin, Austin, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology Virginia, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No